CLINICAL TRIAL: NCT01345760
Title: Expression Levels of RNA-induced Silencing Complex (RISC) Components TARBP1, TARBP2, Argonaute-1, Argonaute-2, PACT and Microprocessor Complex Component DGCR8 in Epithelial Skin Cancer
Brief Title: Expression Levels of RISC and Microprocessor Complex Components in Epithelial Skin Cancer
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Dr., Ruhr University of Bochum
Other Study IDs: 1-Sand
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Skin Cancer
Keywords: Basal Cell Carcinoma; Squamous Cell Carcinoma; Actinic Keratosis; microRNA; Dicer; Drosha; RISC; microprocessor complex; Argonaute; DGCR8; TARBP
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Keratosis, Actinic; Rhabdomyosarcoma, Embryonal, 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — human skin
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Basal Cell Carcinoma
- Squamous Cell Carcinoma
- Actinic Keratosis
- healthy non-lesional skin

SUMMARY:
MicroRNAs (miRNAs) are very small endogenous RNA molecules about 22-25 nucleotides in length, capable of post-transcriptional gene regulation. miRNAs bind to their target messenger RNAs (mRNAs), leading to cleavage or suppression of target mRNA translation based on the degree of complementarity. miRNAs have recently been shown to play pivotal roles in diverse developmental and cellular processes and linked to a variety of skin diseases and cancers. In the present study, the investigators examines the expression profiles of the microprocessor complex subunit DGCR8 and the RISC components TARBP1, TARBP2, argonaute-1, argonaute-2 and PACT in epithelial skin cancer and its premalignant stage.

DETAILED DESCRIPTION:
Patients with premalignant actinic keratoses, basal cell carcinomas and squamous cell carcinomas were included in the study. Punch biopsies were harvested from the center of the tumors, from sites of healthy skin and a healthy control group. DGCR8, TARBP1, TARBP2, argonaute-1, argonaute-2 and PACT mRNA expression levels were detected by quantitative real-time reverse transcriptase polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* epithelial skin cancer

Exclusion Criteria:

* other known previous malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial skin cancer and pre-malignant stages
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Falk G Bechara, PD Dr., Study Director — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum
Locations (1):
- Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Skrygan M, Georgas D, Arenz C, Gambichler T, Sand D, Altmeyer P, Bechara FG. Expression levels of the microRNA maturing microprocessor complex component DGCR8 and the RNA-induced silencing complex (RISC) components argonaute-1, argonaute-2, PACT, TARBP1, and TARBP2 in epithelial skin cancer. Mol Carcinog. 2012 Nov;51(11):916-22. doi: 10.1002/mc.20861. Epub 2011 Oct 24. PMID 22025453